CLINICAL TRIAL: NCT02690298
Title: Evaluation of ExSpiron™ Non-Invasive Respiratory Volume Monitor Measurements Derived Without Patient Specific Calibration
Brief Title: Evaluation of ExSpiron™ Measurements Derived Without Patient Specific Calibration
Acronym: RMI UVU
Status: Completed | Type: Observational
Sponsor: Respiratory Motion, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RMI UVU 2015-0052
Record Dates: First submitted 2015-09-08; First posted 2016-02-24 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Non-Invasive Respiratory Volume Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: ExSpiron — Non-Invasive respiratory volume monitoring
  Other Names: RVM

SUMMARY:
Previous studies have shown that the ExSpiron™ can provide non-invasive, real-time, accurate measurements of minute ventilation (MV), tidal volume (TV) and respiratory rate (RR) after calibration with a spirometer. The purpose of this study is to compare the MV, TV and RR values measured by the ExSpiron™ without prior spirometer calibration to values obtained with a spirometer calibration. In this study, the MV and TV values will be compared between the ExSpiron™ with and without prior patient-specific calibration of the ExSpiron™ to a spirometer

DETAILED DESCRIPTION:
In order to evaluate the performance of the device under the range of conditions encountered in the clinical environment, the respiratory volume monitor (RVM) was tested throughout a range of respiratory rates and also during erratic breathing patterns. At 4 and 36 breaths per minute (the extremes of the rates anticipated to be encountered in the clinical setting), and during erratic breathing, RVM and spirometry measurements were found to be highly-correlated (r=0.98 ±0.01 (mean ±95%CI) at 4 breaths/min, 0.97 ±0.01 at 36, and 0.93 ±0.04 during erratic breathing). These studies also included calibration of the ExSpiron to the spirometer.

The primary objective of the study is to compare the minute ventilation (MV), tidal volume (TV) and respiratory rate (RR) measurements collected and reported by the ExSpiron, without prior ExSpiron calibration, against acquired MV, TV, and RR measurements from an ExSpiron with prior individual specific calibration to a spirometer using either a Wright Spirometer or a Morgan Flow Volume Loop (FVL) Pneumotachograph Spirometer. A secondary objective will be to confirm the PadSet functionality after 24 hours of wear in accordance with current labeling.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females aged 21-90
* Able to provide written informed consent
* Able to participate in a two day study

Exclusion Criteria:

* Men and Women aged <21 years and >90 years of age
* Inability to follow study and/or study staff instructions
* Inability to perform study procedures, e.g. spirometry
* Allergy to the electrodes or components of the electrodes

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Respiratory measurements will be acquired from up to 100 subjects from a wide cross-section of the adult population. Potential subjects will be screened based on the following inclusion/exclusion criteria to determine eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure of the study is the minute ventilation (MV), in liters per minute (L/min), collected and reported by the ExSpiron, with and without prior ExSpiron calibration | 3 months
  Calibrated ExSpiron measurements compared against uncalibrated ExSpiron measurements
The primary outcome measure of the study is the tidal volume (TV), in liters (L), collected and reported by the ExSpiron, with and without prior ExSpiron calibration | 3 months
  Calibrated ExSpiron measurements compared against uncalibrated ExSpiron measurements
The primary outcome measure of the study is the respiratory rate (RR), in breaths per minute (bpm), collected and reported by the ExSpiron, with and without prior ExSpiron calibration | 3 months
  Calibrated ExSpiron measurements compared against uncalibrated ExSpiron measurements